CLINICAL TRIAL: NCT01596725
Title: A Phase 1 Randomized, Observer-Blinded, Dose-Ranging Study to Evaluate the Immunogenicity and Safety of Monovalent A/Indonesia/05/05 (H5N1) Virus-Like Particle (VLP) Avian Influenza Antigen (Recombinant) in Healthy Young Adults With and Without Adjuvant 2.
Brief Title: A/H5N1 Virus-Like Particle Antigen Dose Ranging Study With Adjuvant 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novavax (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NVX778.P102
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Influenza (Pandemic)
MeSH Terms: conditions — Influenza, Human | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group A (Experimental)
  Interventions: Biological: Monovalent Avian Influenza VLP (H5N1)
- Group B (Experimental)
  Interventions: Biological: Monovalent Avian Influenza VLP (H5N1)
- Group C (Experimental)
  Interventions: Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant
- Group D (Experimental)
  Interventions: Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant
- Group E (Experimental)
  Interventions: Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant
- Group F (Experimental)
  Interventions: Biological: Saline Placebo

INTERVENTIONS:
Biological: Monovalent Avian Influenza VLP (H5N1) — Dose A without Adjuvant 2; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group A
Biological: Monovalent Avian Influenza VLP (H5N1) — Dose B without Adjuvant 2; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group B
Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant — Dose B with Adjuvant 2; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group C
Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant — Dose C with Adjuvant 2; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group D
Biological: Monovalent Avian Influenza VLP (H5N1); Adjuvant — Dose D with Adjuvant 2; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group E
Biological: Saline Placebo — Placebo; intramuscular, deltoid, Day 0 and Day 21
  Arms: Group F

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety profile of the Avian flu vaccine with and without adjuvant 2 in healthy, young adults. The study is divided down into Parts A1, A2 and B. Groups within each Part will receive two doses of the assigned test article on Study Days 0 and 21. There will be a Safety Monitoring Committee assessment following Day 7 for each part, prior to allowing vaccination of subjects in subsequent Parts of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female, ≥18 and ≤49 years of age,
2. Willing and able to give informed consent prior to study enrollment,
3. Able to comply with study requirements, and
4. All women must have a negative urine pregnancy test prior to each vaccination. Women will be advised through the Informed Consent process to avoid becoming pregnant over the duration of the study, and must assert that they will employ an effective form of birth control for the duration of the study. Acceptable forms of birth control are: credible history of abstinence from heterosexual activity or prior surgical sterilization, hormonal contraceptives (oral, injectable, implant, patch, ring), double-barrier contraceptives (condom or diaphragm, with spermicide), and intrauterine device (IUD).

Exclusion Criteria:

1. Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care. Asymptomatic conditions (e.g., hypertension, dyslipidemia) that are being managed medically and that are not associated with evidence of end-organ damage are not exclusionary provided they are clinically stable (defined as no unscheduled medical interventions or change in medications for cause within 3 months).
2. Any history of jaundice, or of hepatic injury due to drug (prescription, OTC, or illicit) or alcohol use or viral hepatitis; or the presence of hepatitis B surface antigen or hepatitis C antibody at screening.
3. Any grade 1 or higher (as based on the Toxicity Grading Scale [TGS]) abnormality in serum glutamic-pyruvic transaminase/alanine aminotransferase (SGPT/ALT), serum glutamic-oxaloacetic transaminase/aspartate aminotransferase (SGOT/AST), alkaline phosphatase, or total bilirubin levels.
4. Any grade 2 or higher (as based on the TGS) vital sign or clinical laboratory abnormality not specified in criterion 3 above. Note that any abnormal vital sign may be repeated at the Investigator's discretion.
5. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination.
6. History of a serious reaction to prior influenza vaccination.
7. History of Guillain-Barré Syndrome (GBS) within 6 weeks following a previous influenza vaccine.
8. Received any vaccine in the 4 weeks preceding the study vaccination; or any A/H5N1 avian influenza vaccine at any time.
9. Any known or suspected immunosuppressive condition, acquired or congenital, including HIV infection, as determined by history and/or physical examination.
10. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10 mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
11. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
12. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature >38.0°C on the planned day of vaccine administration).
13. Known disturbance of coagulation.
14. Women who are pregnant or breastfeeding, or plan to become pregnant during the study.
15. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
16. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic or psychiatric conditions deemed likely to impair the quality of safety reporting).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of solicited and unsolicited adverse events in H5N1 VLP antigen dose groups delivering HA with/without Adjuvant 2. | Day 42

SECONDARY OUTCOMES:
Measurement of HAI antibody seroconversion rates and GMT achieved by a constant H5N1 VLP antigen dose alone and in combination with Adjuvant 2. | Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Thomas, Ph.D, Study Director — Novavax
Locations (5):
- United States (5):
  - Anaheim Clinical Trials, Anaheim, California
  - Miami Research Associates, Miami, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Clinical Trials of Texas, San Antonio, Texas

REFERENCES:
- See also: Related Info — http://www.novavax.com